CLINICAL TRIAL: NCT04097860
Title: Improving Lactation Success in Mothers of Critically Infants Using Personalized Real-Time Biomarker Based Text Messages
Brief Title: Improving Lactation Success in Mothers of Critically Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB201902053
Record Dates: First submitted 2019-09-19; First posted 2019-09-20 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2024-11

CONDITIONS: Breast Pumping
MeSH Terms: conditions — Breast Milk Expression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Individuals monitoring breast milk production and sodium levels will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Will be sent one message that includes general information pertinent to all mothers expressing BM for their infants and one personalized real-time biomarker based message which will include the sodium level contained in the BM since the previous message, the number of times pumped on those days and will either congratulate the participant on how well the is pumping BM for the infant or how many more times per day the participant needs to pump to decrease the BM sodium level and increase BM production
  Interventions: Behavioral: Text message including biomarker of breast pumping adequacy
- Control group (No Intervention): Will only be sent text messages that include the same general lactation information sent to the treatment group

INTERVENTIONS:
Behavioral: Text message including biomarker of breast pumping adequacy — The intervention group will be sent one message that includes general information pertinent to all mothers expressing BM for their infants and one personalized real-time biomarker based message which will include the sodium level contained in the BM since the previous message, the number of times pumped on those days and will either congratulate the participant on how well the participant is pumping BM for the infant or how many more times per day the participant needs to pump to decrease the BM sodium level and increase BM production
  Arms: Intervention group

SUMMARY:
The purpose of this study is to determine the feasibility and potential benefits of a mHealth intervention to increase BM pumping frequency and BM production in mothers delivering critically ill infants admitted to the neonatal intensive care unit

DETAILED DESCRIPTION:
Although compelling evidence exists that breast milk (BM) improves infant health, mothers of critically ill infants frequently produce insufficient amounts BM which is likely due to inadequate daily breast pumping frequency. BM sodium levels are an easy to measure biomarker of pumping frequency and providing this information to mothers via text messaging may increase their pumping frequency and BM production. Therefore, the overall objective of this pilot study is to determine the feasibility and potential benefits of a mHealth intervention to increase BM pumping frequency and BM production in mothers delivering critically ill infants admitted to the neonatal intensive care unit (NICU) at University of Florida Health. Specific aims include (1) evaluate the feasibility of a mHealth intervention to increase BM pumping frequency and BM production and (2) assess whether results indicate a signal of effectiveness supporting a subsequent adequately powered randomized clinical trial (RCT). Following delivery, 50 mothers of critically ill infants admitted to the NICU will be randomized to one of two groups. The Enhanced Intervention Group will receive text messages including both general lactation information and a personalized message consisting of the mother's BM sodium level, pumping frequency and feedback regarding pumping frequency. The Standard Intervention Group will receive only general lactation information. Results will be used to revise the intervention and study processes and to estimate outcome measurement variability and effect sizes needed for sample size calculations for an adequately powered RCT.

ELIGIBILITY:
Inclusion Criteria:

* stated intent to provide BM to the infant
* infant not expected to be stable enough to bottle/breastfeed for > 14 days
* owns a mobile phone with unrestricted SMS capability.
* English speaking

Exclusion Criteria:

* known illicit drug use
* breast reduction or augmentation
* positive HIV status
* does not anticipate being able to bring BM to the NICU at least 4X/week
* infant not expected to live > 7 days following delivery
* COVID-19 positive

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2025-09-03 (Actual); Study Completion 2025-09-03 (Actual)

PRIMARY OUTCOMES:
Volume of breast milk (BM) | Up to 2 weeks
  All BM will be weighed (1 mg of BM = 1 mL) by a BM technician and the weight recorded in the infant's medical record. BM will be weighed on a portable digital scale accurate to within 0.1 grams.

SECONDARY OUTCOMES:
Number of breast pumping episodes | Up to 2 weeks
  Daily number of pumping sessions as recorded in the mother's log book and verified by examination of the date and time on vials of pumped BM.
Breast milk sodium level | Up to 2 weeks
  Daily BM sodium levels beginning when the mother has produced at least 5mL of BM and continuing for the two week study.

CONTACTS AND LOCATIONS:
Overall Officials: Leslie A Parker, MD, Principal Investigator — University of Florida
Locations (1):
- UF Health Children's Hospital, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No